CLINICAL TRIAL: NCT05274113
Title: Efficacy of Direct Versus Peripheral Low-Dose Adjuvant Dexamethasone on Duration and Rebound Pain in Regional Anesthesia for Distal Radius Fracture Fixation: A Prospective Randomized Controlled Blinded Study
Brief Title: Low Dose Dexamethasone for Distal Radius Fractures
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MWAN22D.110
Record Dates: First submitted 2022-03-02; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Post Operative Pain; Distal Radius Fracture
MeSH Terms: conditions — Pain, Postoperative; Wrist Fractures | interventions — Dexamethasone; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Block with Ropivacaine + Dexamethasone (Active Comparator): Before surgery an ultrasound guided supraclavicular block with ropivacaine and 4 mg of dexamethasone will be administered
  Interventions: Drug: Dexamethasone 4mg; Drug: Ropivacaine
- Group 2: Ropivacaine Block + IV Dexamethasone (Active Comparator): Before surgery an ultrasound guided supraclavicular block with ropivacaine will be administered and patients will receive dexamethasone intravenously
  Interventions: Drug: Dexamethasone 4mg; Drug: Ropivacaine

INTERVENTIONS:
Drug: Dexamethasone 4mg — 4 mg of Dexamethasone will be given before surgery
Drug: Ropivacaine — Ultrasound guided supraclavicular block with ropivacaine will be given to patients before surgery

SUMMARY:
The addition of the steroid dexamethasone to a single injection of local anesthetic has been shown to significantly prolong the duration of peripheral nerve blockade compared to local anesthetic alone. This allows for improved post-operative pain scores and reduces opioid use in the early post-operative period. However, the use of a steroid adjuvant in regional nerve blocks is generally not considered standard of care, and there is considerable variation among anesthesiologists regarding preferred formulations and the role of adjuvants in regional anesthesia. A recent study from our institution demonstrated the effectiveness of dexamethasone directly mixed with local anesthetic at multiple doses compared to placebo for upper extremity surgery. With this prospective randomized controlled blinded trial, we hope to definitively establish which method of adjuvant dexamethasone administration is superior in extending the effects of a brachial plexus nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 undergoing open reduction and internal fixation of a distal radius fracture less than 3 weeks from injury with a volar plate technique
* American Society of Anesthesiologists (ASA) levels 1 through 3 at time of surgery
* Opioid naïve patients

Exclusion Criteria:

* History of Drug/opioid/alcohol abuse
* Polytrauma patients
* History of inflammatory disorder, infection, dementia, psychiatric/neurological disorder, relevant drug/local anesthesia allergy, relevant chronic upper extremity pain (RSD, fibromyalgia, neuralgia, etc)
* Excessive BMI
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-10 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain control | 72 hours
  Measured using participants Visual Analog Scale (VAS) pain scores
Postoperative pain control #2 questionnaire | 72 hours
  Measured by asking participants how much medication they take after surgery to help control their pain

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States